CLINICAL TRIAL: NCT06588933
Title: The Development and Validation of a Novel Tool for the Assessment of Taste Disturbances in Patients With Advanced Cancer: Taste Questionnaire in Palliative Care
Brief Title: TQ-PAL Development and Validation
Status: Recruiting | Type: Observational
Sponsor: Prof Andrew Davies (Other)
Responsible Party: Sponsor-Investigator, Prof Andrew Davies, Professor of Palliative Medicine, Our Lady's Hospice and Care Services
Organization: Our Lady's Hospice and Care Services (Other)
Other Study IDs: Our Lady's Hospice
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Altered Taste
Keywords: neoplasm
MeSH Terms: conditions — Dysgeusia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: completion of a questionnaire — completion of a questionnaire by participant

SUMMARY:
Taste problems are common among patients with advanced cancer. These symptoms can affect the pleasure of eating and drinking, reduce dietary intake, cause low mood, and a lower quality of life. There is no validated tool to assess taste disturbances and their impact on patients with advanced cancer. This study will develop and validate a novel assessment tool to assess taste disturbances and their impact on patients with advanced cancer.

DETAILED DESCRIPTION:
Patients with advanced cancer often develop taste disturbances. A recent literature review reported a median prevalence of 55%, with prevalence ranging from 27-93%. Studies have shown taste disturbance is usually a persistent symptom, is often 'moderate-to-severe' in intensity, and is often associated with significant distress. Taste disturbance may have a major impact on the experience and pleasure associated with eating and drinking. Taste disturbance may have a major impact on nutritional intake. It may be associated with low mood / depression, social isolation, and an impaired quality of life.

The aforementioned literature review identified, importantly, that the terminology used in the published literature varied, which may have had an effect on the results obtained, especially prevalence statistics. The review identified the need for "development/validation studies of a taste-specific assessment tool for this group of patients - there is a need for a tool that not only assesses the problem but can also assess the response to treatment for the problem, utilising patient reported outcome measures."

ELIGIBILITY:
Inclusion Criteria:

18 years of age Diagnosis of locally advanced or metastatic cancer Referred to palliative care/oncology services Taste problems rated 'moderate' or worse over previous 2-week period Good understanding of English

Exclusion Criteria:

Cognitive impairment (unable to provide consent / complete questionnaire) Taste problems precedes cancer diagnosis. Head and neck surgery Head and neck radiotherapy Salivary gland disorders (e.g., Sjogren's Syndrome) In the 'Deteriorating' or 'Terminal' Phase of illness

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are currently under the care of oncology or palliative care who have an incurable cancer. Patients will be identified by the clinical teams at the study sites, informed about the study, and (if interested in taking part in the study) referred to the research team. Participants will be screened for inclusion by asking 1. Over the past 2 weeks have you experienced taste problems?" If yes to the question, "How severe was it? (Options- Slight/Moderate/Severe/Very severe)". Patients must score as moderate/severe/very severe
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To develop a novel assessment tool to assess taste disturbances in patients with advanced cancer | December 2025
  To develop the Taste Questionnaire in Palliative Care (TQ-PAL) to assess taste disturbances and their impact on patients with palliative care. It's domains include the effect on food intake, social inclusion, and quality of life
To validate the newly developed Taste Questionnaire in Palliative Care (TQ-PAL) | December 2025
  To test the TQ-PAL for face, content, construct, convergent and reliability validation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, FRCP, Principal Investigator — Our Lady's Hospice and Care Services
Locations (1):
- Our Lady's Hospice & Care Services, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hannon M, Shaw A, Connolly M, Davies A. Taste disturbance in patients with advanced cancer: a scoping review of clinical features and complications. Support Care Cancer. 2023 Sep 6;31(10):562. doi: 10.1007/s00520-023-08012-x. PMID 37672147
- [Background] McGettigan N, Dhuibhir PU, Barrett M, Sui J, Balding L, Higgins S, O'Leary N, Kennedy A, Walsh D. Subjective and Objective Assessment of Taste and Smell Sensation in Advanced Cancer. Am J Hosp Palliat Care. 2019 Aug;36(8):688-696. doi: 10.1177/1049909119832836. Epub 2019 Mar 3. PMID 30827119
- [Background] Hutton JL, Baracos VE, Wismer WV. Chemosensory dysfunction is a primary factor in the evolution of declining nutritional status and quality of life in patients with advanced cancer. J Pain Symptom Manage. 2007 Feb;33(2):156-65. doi: 10.1016/j.jpainsymman.2006.07.017. PMID 17280921
- [Background] Kirkova J, Walsh D, Rybicki L, Davis MP, Aktas A, Tao Jin, Homsi J. Symptom severity and distress in advanced cancer. Palliat Med. 2010 Apr;24(3):330-9. doi: 10.1177/0269216309356380. Epub 2009 Dec 16. PMID 20015920